CLINICAL TRIAL: NCT02025946
Title: Observational Study of Total Ankle Arthroplasty and Tibiotalar Arthrodesis
Status: Withdrawn | Type: Observational
Sponsor: Integra LifeSciences Services (Industry)
Responsible Party: Sponsor
Other Study IDs: RECON-EMEA-12
Record Dates: First submitted 2013-12-31; First posted 2014-01-01 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Total Ankle Arthroplasty
- Tibiotalar Arthrodesis

SUMMARY:
In case of severe ankle arthritis, the two common surgical treatments are tibiotalar arthrodesis and total ankle arthroplasty. Few studies have compared these treatments and it remains difficult to determine which operation is the better solution for end stage ankle arthritis.

The purpose of the present study is to analyze patient's outcome after each type of ankle surgery and to describe the decision making process.

ELIGIBILITY:
Inclusion Criteria:

* Patient with isolated symptomatic end-stage ankle arthritis who needs a tibiotalar arthrodesis or a mobile-bearing total ankle arthroplasty
* Patient receiving CE marked medical devices and planned to be operated in compliance with their respective Instructions for Use
* Patient aged between 40 and 75 years old

Exclusion Criteria:

* Patient who already had before his inclusion in this study a tibiotalar arthrodesis or a total ankle arthroplasty in the same ankle
* Patient with planned or existing arthrodesis of adjacent joints (subtalar, talonavicular and calcaneaocuboid joint)
* Patient with ankle deformity > 20° (weight bearing X-rays)
* Patient with history of infection of the ankle joint (positive culture) or current infection of the ankle joint (positive culture)
* Patient with neuropathy or with a history of diabetes mellitus for more than 15 years
* Patient with avascular necrosis of the talus >25%
* Patient already included in the study for the other ankle

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with isolated symptomatic end-stage ankle arthritis who needs a tibiotalar arthrodesis or a mobile-bearing total ankle arthroplasty, receiving CE-marked medical devices and planned to be operated in compliance with their respective Instructions for Use
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2021-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
proportion of reoperations in the total ankle replacement arm and in the tibiotalar arthrodesis arm | after 5 years of follow-up
  Reoperation will be defined as any secondary surgery related to the operated ankle or adjacent joints (subtalar, talonavicular and calcaneocuboid joints), excluding wound healing problems.

SECONDARY OUTCOMES:
Proportion of reoperation in the tibiotalar arthrodesis arm and in the total ankle replacement arm | 1, 2, 7 and 10 years
  The proportion of reoperation as defined above and for the whole study period in the tibiotalar arthrodesis arm and in the total ankle replacement arm
proportion of revision for the whole study period in the tibiotalar arthrodesis arm and in the total ankle replacement arm | 1, 2, 5, 7 and 10 years
  For the arthrodesis arm, a revision will be defined as a reoperation for one of the following reasons: nonunion or pseudoarthrosis or malunion. Hardware removal will not be considered as a revision.
  For the total ankle arthroplasty arm, a revision will be defined as the change of any metallic component of the implanted device. The incidental change of the polyethylene will not be considered as a revision except when it is broken without any
The evolution and clinical outcomes | 1, 2, 5, 7 and 10 years
  * Pain measured using a Visual Analog Scale (VAS)
  * Ankle function measured using the American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Scale
  * Level of activity measured using the University of California, Los Angeles (UCLA) activity scale
  * Quality of life measured using the EQ5D™ questionnaire
  * Arthritis status of adjacent joints measured using the Kellgren-Lawrence grading scale
  * Patient satisfaction
the decision criteria for choosing the surgical technique use | inclusion
  Reason for choosing the Total ANkle Arthroplasty or Tibiotalar Arthrodesis

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen De Wachter, Principal Investigator — AZ Turnhout
Locations (8):
- Belgium (2):
  - Katholieke Universiteit Leuven, Leuven
  - AZ Turnout - Clinic Sint-Jozef, Turnhout
- Clinique Axium, Aix-en-Provence, France
- I.R.C.C.S. Istituto Ortopedico Galeazzi, Milan, Italy
- Sint Lucas Andreas Ziekenhuis, Amsterdam, Netherlands
- Hospital Pedro Hispano, Matosinhos Municipality, Portugal
- Hospital clinico y provincial, Barcelona, Spain
- Musgrave Park Hospital, Belfast, United Kingdom